CLINICAL TRIAL: NCT03288441
Title: Management Patterns of AntiThrombotics and Outcomes in Patients With Hematological Malignancy and ThrombocytopEnia: a Prospective Registry (MATTER Study)
Brief Title: Management and Outcomes of Anti-thrombotic Medication Use in Thrombocytopenia
Acronym: MATTER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: METC 17-4-061
Record Dates: First submitted 2017-09-07; First posted 2017-09-20 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Hematologic Neoplasms; Thrombocytopenia; Anticoagulants; Platelet Aggregation Inhibitors
Keywords: Hematologic Neoplasms; Thrombocytopenia; Anticoagulants; Platelet Aggregation Inhibitors
MeSH Terms: conditions — Hematologic Neoplasms; Thrombocytopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — After measuring the activity of anticoagulant drugs from the plasma when doses are modified, remaining plasma will be retained for 5 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- antiplatelet only: Patients receiving antiplatelet medication, but not anticoagulation. Antiplatelet drugs include any class, dose or duration of any platelet aggregation inhibitor.
  This refers to the antithrombotic regimen when the current thrombocytopenia, or risk thereof (i.e. "predicted"), was first identified (even if the treatment is subsequently stopped)
  Interventions: Drug: Hold; Drug: Change antithrombotic Drug; Biological: Change platelet transfusion threshold; Drug: Full dose antithrombotics
- anticoagulant-based: Patients receiving only anticoagulants or both anticoagulant and antiplatelet medication combined. This includes any class, dose or duration of any antiplatelet or anticoagulant drug.
  This refers to the antithrombotic regimen when the current thrombocytopenia, or risk thereof (i.e. "predicted"), was first identified (even if the treatment is subsequently stopped)
  Interventions: Drug: Hold; Drug: Prophylactic dose antithrombotic; Drug: Change antithrombotic Drug; Biological: Change platelet transfusion threshold; Drug: Full dose antithrombotics; Device: Mechanical measures; Drug: Intermediate dose antithrombotic

INTERVENTIONS:
Drug: Hold — Hold antithrombotic therapy
Drug: Prophylactic dose antithrombotic — Reduction in antithrombotic medication dose to prophylactic dose (without changing type)
  Groups: anticoagulant-based
Drug: Change antithrombotic Drug — Change in type of antithrombotic therapy
Biological: Change platelet transfusion threshold — Increase or reduce platelet transfusion threshold
Drug: Full dose antithrombotics — Continue full dose antithrombotic therapy
Device: Mechanical measures — Mechanical measures to reduce thrombotic risk including: IVC filter insertion, Intermittent Pneumatic Compression (IPC), Removal of Central venous catheter
  Groups: anticoagulant-based
Drug: Intermediate dose antithrombotic — Reduction in antithrombotic medication dose to prophylactic dose (without changing type). Intermediate dose in between prophylactic and full dose
  Groups: anticoagulant-based

SUMMARY:
Background: Antithrombotic therapy in the context of treatment related thrombocytopenia (i.e. low levels of platelets) is not uncommon. Guidelines are based upon a paucity of retrospective data and focus on the scenario of cancer associated venous thrombosis and low molecular weight heparin treatment. Even less is known regarding direct oral anticoagulants, antiplatelet therapy, or anticoagulation prescribed for other indications.

Aims: The study aims are to evaluate how physicians manage anticoagulant and antiplatelet medication in patients with hematological malignancy and thrombocytopenia, and to assess the frequency of bleeding and thrombosis. Additional aims are to assess how management changes affect drug activity and blood clotting (coagulation), and to evaluate the use of platelet transfusions.

Design: The investigators plan a multinational prospective registry of patients admitted to the inpatient hematology department or outpatient clinic at one of the study centers. Patients with hematological malignancies, platelets below 50 X 109/L, and anticoagulant and/or antiplatelet medication will be studied.

Patients will be enrolled when the combination of antiplatelet/anticoagulant medication and thrombocytopenia is first detected. Patients will be followed until 30 days after the baseline study visit (which occurs 30 days after enrollment or when platelets < 50*109/L, whichever come first) or death. Patients will be indexed at the time of baseline visit.

Patients will be excluded from study analysis if one of the following events occurs before study index: Withdrawal of consent, death, clinically-relevant non-major bleeding or the composite primary outcome.

Risk factors for bleeding and thrombosis will be recorded at baseline. Parameters from routine blood tests will be recorded throughout the study. During the study major bleeding events and thrombosis will be recorded. Investigational blood tests assessing coagulation and drug activity will be drawn at baseline (=study index). Throughout the study all management decisions regarding antithrombotic therapy, including platelet and red blood cell transfusion, will be recorded. This is an observational study and management will be solely at the discretion of the physician.

Analysis: The investigators will first look at the frequency of either bleeding or thrombosis according to the type of management strategy and evaluate the platelet threshold at which a given management strategy is employed.

At the next stage, in selected subgroups, the optimal management strategy with respect to bleeding/thrombotic risk, will be determined.

DETAILED DESCRIPTION:
* Thrombocyte-level cohorts Patients will be divided into two groups based on the platelet level at study index .

  1. Thrombocytopenic Cohort: Patients with morning platelet count below 50*109/L at study index. This is the main study cohort for all analyses
  2. Non-thrombocytopenic Cohort: Patients whose morning platelet count is ≥ 50*109/L at study index will be considered as a reference group, and not included in the primary analysis.
* Analysis of outcomes:

By definition, there will be an intervention at the time of study index (baseline), meaning that even if no change is made, it will be considered an intervention. Each patient may have multiple exposures/interventions over the study.

Therefore, in a time dependent analysis, each outcome will be linked to the exposure/intervention at study index.

Each exposure/intervention will be linked with the platelet level on the day of the intervention.

#Competing Events:

The following events (in addition to death) will be considered competing events and will be considered as such in the statistical analyses of the outcomes:

1. The composite primary outcome
2. change in the antithrombotic regimen after study index
3. diagnosis of HIT or TTP
4. a change in the hematological malignancy treatment regimen. Study follow-up will continue after these events, and study data will continue to be recorded until censorship for end of study period or death.

   * Detecting selection bias:

Patients fulfilling the inclusion criteria but not included in the study, will be detected by reviewing the medical records of the hematology institute, weekly. The baseline characteristics and reason for not including these patients will be recorded retrospectively in the "not-included cohort". The baseline characteristics of this cohort will be compared with the study cohort to ascertain whether selection bias exists.

ELIGIBILITY:
Inclusion Criteria:

* Any hematological malignancy with or without active treatment (including autologous or allogeneic stem cell transplantation), irrespective of the treatment line and disease status.
* Disease-related and/or current/predicted treatment-related thrombocytopenia (<50 X 109/L) of any duration.
* Current antiplatelet and/or anticoagulant treatment of any duration and for any indication. This treatment may have been started before or after diagnosis of the hematological malignancy and thrombocytopenia.

"Current" refers to the time when the current thrombocytopenia, or risk thereof (i.e. "predicted"), was first identified (even if the treatment is subsequently stopped)

Exclusion Criteria:

* Previous thrombocytopenia (<50 X 109/L) while using the current antithrombotic regimen.
* Current diagnosis of heparin induced thrombocytopenia (HIT) or thrombotic thrombocytopenia purpura (TTP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects treated at the inpatient or outpatient hematology departments at the participating centers
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-03-20 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite of major bleeding or thrombosis | 30 days (from study index) or until death (whichever first)
  1) ISTH-defined Major bleeding events defined as: Fatal bleeding; bleeding into a critical organ; clinically overt bleeding associated with a decrease in hemoglobin level of more than 2 g/dL or leading to the transfusion of two or more units of blood OR: 2) Thrombosis defined as: Any symptomatic deep or superficial venous or arterial thromboembolism demonstrated on objective imaging/laboratory tests. Ischemic strokes with no immediate imaging signs will also be considered events, provided this was diagnosed by a neurologist and that the patient had objective neurological signs.

SECONDARY OUTCOMES:
Platelet transfusion related adverse effects | 30 days (from study index) or until death (whichever first)
  Number of adverse effects (all types and individually grouped) related to platelet/plasma transfusion, occurring within 24 hours of transfusion
Clinically Relevant non-Major Bleeding | 30 days (from study index) or until death (whichever first)
  Defined according to the ISTH criteria published in the journal of thrombosis and Hemostasis by Kaatz et al in 2015
Number of platelet tranfusions | 30 days (from study index) or until death (whichever first)
  Number of platelet transfusions
Number of RBC tranfusions | 30 days (from study index) or until death (whichever first)
  Number of red blood cell transfusions
Death | 30 days (from study index)
  death from any cause
Change in antithrombotic management | 30 days (from study index) or until death (whichever first)
  Change in dose/type of antiplatelet or anticoagulant medication OR change in platelet threshold, AFTER the initial intervention which was recorded at study index.

OTHER OUTCOMES:
peak anticoagulant intensity | 3 days after study index
  anti-Xa, Hemoclot, INR, aPTT will be measured at peak, depending on the anticoagulant drug. Patients will be classified as having sub-therapeutic, therapeutic, supra-therapeutic treatment levels, based upon the reference range at the central laboratory. Only relevant for patients with anticoagulation undergoing dose change.
Whole blood coagulation | 3 days after study index
  Measured by rotational thromboelastometry (ROTEM) drawn at study index

CONTACTS AND LOCATIONS:
Overall Officials: Avi Leader, MD, Principal Investigator — Rabin Medical Center, Petah Tikva, Israel; Hugo ten Cate, MD, PhD, Study Chair — Maastricht University Medical Center, Maastricht; Anna Falanga, MD, Study Chair — A.O. Papa Giovanni XXIII - S.I.M.T.
Locations (21):
- Oregon Health & Science University Hospital, Portland, Oregon, United States
- Israel (4):
  - Rambam Health Care Campus, Haifa
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (11):
  - Azienda Ospedaliera Nazionale SS. Antonio e Biagio e C. Arrigo di Alessandria, Alessandria
  - A.O. Papa Giovanni XXIII - S.I.M.T., Bergamo
  - ASST degli Spedali Civili di Brescia, Brescia
  - A.O.U. di Modena, Modena
  - Ospedale San Gerardo di Monza, Monza
  - University Hospital Policlinico di Palermo, Palermo
  - A.O.U Policlinico Umberto I di Roma, Roma
  - Fondazione Policlinico Universitario A. Gemelli, Roma
  - Università degli studi di Roma "Tor Vergata", Roma
  - A.O.U. CITTA' della SALUTE e della SCIENZA di TORINO, Torino
  - AZIENDA ULSS N. 8 BERICA di Vicenza, Vicenza
- Netherlands (5):
  - Amsterdam University Medical Centers, Amsterdam
  - University Medical Center Groningen, Groningen
  - Maastricht University Medical Center (MUMC+), Maastricht
  - Erasmus Medical Center, Rotterdam
  - HagaZiekenhuis, The Hague